CLINICAL TRIAL: NCT05233228
Title: Mobile Health Technology for Personalized Tobacco Cessation Support in Laos
Acronym: SupportLaos
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Setthathirath Hospital (Other); Champasak Hospital, Lao PDR (Unknown); National Center for Laboratory and Epidemiology, Lao PDR (Other); National Tobacco Control Committee, Lao PDR (Other); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12189
Record Dates: First submitted 2022-01-18; First posted 2022-02-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Automated Treatment (Experimental): Consists of all SC components plus a fully automated smartphone-based treatment program that involves interactive and personalized proactive messages, images, or videos.
  Interventions: Drug: Nicotine patch; Behavioral: Self-help materials (to support smoking cessation); Behavioral: Smartphone-based automated treatment for smoking cessation
- Standard Care (Active Comparator): Consists of brief advice to quit smoking delivered by research staff, self-help written materials, and a 2-week supply of nicotine replacement therapy (transdermal patches).
  Interventions: Drug: Nicotine patch; Behavioral: Self-help materials (to support smoking cessation)

INTERVENTIONS:
Drug: Nicotine patch — Provision of nicotine replacement medications in the form of transdermal patches is important to address nicotine withdrawal/craving for smokers who want to quit. Evidence supporting the safety and efficacy of NRT is vast. The PHS Guideline indicates that use of NRT doubles quit rates and should be considered the minimal standard care. Therefore, we will provide NRT to all participants in both groups in the early cessation phase.
Behavioral: Self-help materials (to support smoking cessation) — The self-help materials were developed by NTCC in Lao, based on the World Health Organization's "A guide for tobacco users to quit".
Behavioral: Smartphone-based automated treatment for smoking cessation — The automated treatment(AT) include text messages, images, and videos. The AT content is designed to tap the theoretical mechanisms described in the Phase-Based Model (PBM). That is, treatment content is designed to increase motivation, self-efficacy, use of coping skills, and social support, while reducing nicotine withdrawal symptoms and stress. The AT will begin immediately after enrollment and continue for a 26-week period. The AT approach allows for several levels of personalization for each participant, including tailoring to participants' specific health conditions, individual cessation phases, and participants' self-efficacy level or smoking status in the past week.
  Arms: Automated Treatment

SUMMARY:
In Lao People's Democratic Republic (Lao PDR), 51% of adult men and 7% of adult women smoke tobacco. The development and evaluation of sustainable tobacco cessation interventions suitable for widespread adoption in nations such as Lao PDR are pressing public health needs. To address this need, the investigators propose a project that adapts a theoretically and empirically based mobile health (mHealth) technology to help people quit smoking cigarettes in Lao PDR. This mHealth approach includes a fully automated, interactive, personalized, smartphone-delivered intervention for behavioral treatment, delivered through our Insight™ platform.

This proposed project for Lao PDR includes 2 main phases. In the R21 Phase, the investigators will use formative research methods to adapt our intervention content to the sociocultural context, language, and communication styles of Laotians. In the subsequent R33 Phase, the investigators will conduct a randomized controlled trial (RCT) to evaluate the efficacy of our mHealth intervention and technology. Adult smokers of both sexes will be recruited through 2 large hospitals: Setthathirath Hospital in Vientiane and Champasak Hospital in Champasak Province. Participants (n=500) will be randomized to 1 of 2 treatment groups: Standard Care (SC; n=250) or Automated Treatment (AT; n=250). SC consists of brief advice to quit smoking delivered by research staff, self-help written materials, and a 2-week supply of NRT (transdermal patches). AT consists of all SC components plus a fully automated smartphone-based treatment program that involves interactive and personalized proactive messages, images, or videos. The primary health outcome of the trial is biochemically confirmed self-reported 7-day point prevalence abstinence 12 months post study enrollment. The project also aims to advance mHealth research capacity in Lao PDR and sustain the US-Lao PDR research network. The project has the potential to transform healthcare services for tobacco cessation treatment throughout the country and, ultimately, to reduce tobacco-induced morbidity and mortality significantly.

DETAILED DESCRIPTION:
R21 Phase: Adaption of the AT intervention content

In stage 1, formative research, including literature searches, quantitative results, and qualitative methods (e.g., key informant interviews) are often conducted to determine how well an original intervention will fit the needs and preferences of the target population. The investigators will conduct in-depth interviews with 30 healthcare providers at participating hospitals to learn more about how they typically motivate patients to quit smoking and stay abstinent. Inclusion criteria for all healthcare providers in the R21 Phase include 1) age ≥18 years; and 2) the ability to provide written informed consent to participate. They can develop intervention messages if they wish or pinpoint the sources of treatment content that they use. The investigators will use purposive sampling to select 15 providers from each hospital, 15 of each sex, and ensure the sample is diverse with regard to age and specialty. Also, the investigators will conduct 8 focus group discussions with 40-60 patients who smoke (5-8 persons/group, 4 groups/hospital) to identify additional factors that motivate patients to quit smoking and stay abstinent, barriers to quitting, and strategies to overcome these barriers. Inclusion criteria for all patients in the R21 Phase include 1) age ≥18 years; 2) self-reported current combustible cigarette smoking (smoked ≥100 cigarettes in lifetime and currently smoke ≥1 cigarette/day); 3) planning to quit in the next 6 months or having actually made a quit attempt; and 4) the ability to provide written informed consent to participate. The investigators will use purposive sampling to select a diverse sample with regard to age, residence (urban vs. rural), disease type, and cessation phase, per the Phase-Based Model (PBM; see Conceptual Framework). The investigators will conduct separate group discussions for men and women (2 groups for each sex at each hospital). For all qualitative components in the R21 Phase, the investigators will use open-ended questions in all interviews/discussions. All interviews/discussions will be recorded using a digital voice-recording app on an encrypted smartphone and will be transcribed verbatim. Qualitative data will be analyzed using thematic content analysis with the aid of the R-based Qualitative Data Analysis software package. Themes will be based on the purpose of each component and on theoretical constructs of the PBM.

In stage 2, the investigators will integrate information gathered in the first stage to modify the original intervention. Also at this stage, the investigators will translate all English intervention materials and assessments that will be used in the R33 Phase to Lao, mirroring the WHO's recommended methodology. First, a health scientist, whose native language is Lao, will lead the forward translation process, focusing on conceptual (vs. literal) meaning and comprehensible language for the broadest audience. Second, a more senior bilingual health expert will review the translation, discuss disagreements with the forward translator, edit, and finalize the forward translation. Third, 2 other bilingual health professionals will independently rate the quality of the translation on 5 dimensions: conceptual equivalence, clarity in meaning, comprehensibility, use of common simple language, and cultural appropriateness. Any discrepancies will be discussed to reach consensus on translation or editing. Fourth, the investigators will conduct 6 panel discussions (1 with female smokers, 1 with male smokers, and 1 with mixed-sex healthcare professionals at each participating hospital; 5-7 panelists per group). This step aims to evaluate material comprehensibility as well as linguistic and cultural appropriateness for the target populations, particularly to identify linguistic differences by regions (north vs. south) in Lao PDR and to find and use common words. Fifth, 2 other bilingual health professionals will independently backward translate the materials into English. Finally, the PI and site-PI will independently review and rate the backward-translations for conceptual equivalence with the original English versions.

In stage 3, the investigators will load the intervention content onto the Insight™ platform and assessments into REDCap and will preliminarily test them (on smartphones/ tablets) with 20 patients who smoke (10 male, 10 female). Additionally, the investigators will systematically document continuous feedback from local investigators and staff members who implement stages 2 and 3 for adaption refinement. In stage 4, the investigators will refine the intervention based on the results and feedback from stage 3. Critical changes at this stage (e.g., major deviations from the original intervention) will only be made in consultation with the leadership team.

Stage 5 will be a 3-month pilot efficacy trial with 50 patients. Activities at this stage will mirror the full efficacy trial in the R33 Phase, except that only 50 patients will be recruited and treatment will last 3 months. In addition to the efficacy outcomes, the investigators will collect data for further adaption and refinement.

R33 Phase: Conduct a RCT to evaluate the efficacy of AT:

Sites and participant recruitment: Participants (n=500) will be recruited from the patient populations at Setthathirath Hospital (SH) in Vientiane and Champasak Hospital (CH) in Champasak Province. All non-emergency patients coming to SH and CH first go to a reception desk to receive a queue number and a basic medical form. A flyer that introduces this study will be attached to the basic medical form. Additionally, the investigators will proactively recruit patients at the Respiratory Disease Screening Units (RDSU) and departments/clinics specializing in women's health (e.g., Gynecology, and Breast and Gynecologic Cancer). Due to the national organization and implementation of NCLE's disease control programs, all patients visiting SH or CH with respiratory symptoms are first examined at the RDSU for type of disease, severity, and whether the disease is included in a national disease control program (e.g., tuberculosis or severe acute respiratory syndrome). Patients are then referred to appropriate departments/clinics or disease control units.

Baseline assessment. Enrolled participants will complete a 45-minute tablet-delivered baseline audio computer-assisted self-interview, managed and delivered by REDCap. Research staff will assist participants complete the assessment if needed. Participants will be assigned to a treatment group using a form of adaptive randomization called minimization, this ensures better group balance regarding participant characteristics and does not impose limitations such as empty or near-empty strata. Randomization variables include biological sex, nicotine dependence, and reading level. All participants will complete a brief training session on smartphone use and the Insight™ app. Smartphones will be loaned to participants who need them.

Treatment groups. Standard Care (SC): Participants randomized to SC will receive brief advice to quit smoking delivered by research staff, NTCC's self-help materials (developed based on the WHO's "A guide for tobacco users to quit"), and a 2-week supply of NRT (patches). SC participants will be asked to complete weekly 4-item smartphone-delivered assessments about their diet (see explanation in Measures) for a 6-month period.

Automated Treatment (AT): Participants in the AT group will receive the SC components (except the dietary assessments) plus proactive personalized messages/images/videos for smoking cessation. The AT content is adapted from the team's previous efforts (see Preliminary Studies), is informed by the R21 phase outcomes, and is designed to tap the theoretical mechanisms described in the PBM. That is, AT content is designed to increase motivation, self-efficacy, and use of coping skills, while reducing nicotine withdrawal symptoms and stress. AT will begin immediately after enrollment and continue for a 26-week period (about 2 messages/images/videos per day). The AT approach allows for several levels of personalization for each participant. First, at baseline, participants will be asked several questions about past quit attempts, preferred coping skills, and the presence or fear of specific health conditions. Treatment content tailored to these responses will be automatically delivered throughout the treatment period. Second, there will be different bins of treatment content for different cessation phases to ensure that AT targets critical mechanisms of each participant's PBM phase, which may dynamically change during treatment. Third, participants will be asked to complete brief (4 items) smartphone-delivered assessments during each week of the AT course. These questions will vary depending on each participant's phase (e.g., current level of intrinsic motivation for preparation or maintenance phases or smoking status in the past week and self-efficacy level for all phases). Treatment content (e.g., types and frequencies of messages) for the following week will be based on responses to these weekly assessments and participant phases (e.g., level of self-efficacy or past-week smoking status). Our team's previous work with disadvantaged populations has observed high adherence (76%) with weekly smartphone assessments across a 6-month timeframe.

Participants will be followed up for 12 months but AT and weekly assessments will stop at month 6.

ELIGIBILITY:
Inclusion Criteria: (pilot RCT in the R21 Phase and main RCT in the R33 Phase):

1. aged ≥18 years
2. self-reported current combustible cigarette smokers (smoked at least 100 cigarettes in lifetime and currently smoke ≥1 cigarette/day)
3. willing to set a quit date within 2 weeks of study enrollment
4. able to provide written informed consent to participate
5. able to read Lao (score ≥4 points on the Rapid Estimate of Adult Literacy in Medicine-Short Form).

Exclusion Criteria: (pilot RCT in the R21 Phase and main RCT in the R33 Phase)

1. history of a medical condition that precludes use of NRT
2. ineligibility to participate based on medical or psychiatric conditions diagnosed by a physician/clinician
3. enrollment in another cessation program or current use of other cessation medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Smoking status at 12 months post-enrollment (R33 Phase) | 12 months post enrollment
  The primary outcome is smoking status at 12 months post-enrollment. Abstinence will be defined as biochemically confirmed self-reported 7-day point prevalence abstinence with expired CO <6 ppm.
Smoking status at 3 months post-enrollment (Pilot RCT, R21 Phase) | 3 months post enrollment
  The primary outcome is smoking status at 3 months post-enrollment. Abstinence will be defined as biochemically confirmed self-reported 7-day point prevalence abstinence with expired CO <6 ppm.

SECONDARY OUTCOMES:
Number of cigarettes smoked per day | In-clinic assessments at months 3 and 12
  At the final follow-up (month 3 for the pilot trial and month 12 for the R33 Phase), participants will be asked to self-report their average current numbers of cigarettes smoked per day

CONTACTS AND LOCATIONS:
Overall Officials: Shweta Kulkarni, MS, Study Director — Stephenson Cancer Center, TSET Health Promotion Research Center of OUHSC
Locations (2):
- Laos (2):
  - Champasak Hospital, Champasak
  - Setthathirath Hospital, Vientiane

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be shared upon request, with an established data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After RCT data collection is complete.
Access Criteria: After an institutionally approved data sharing agreement is established, deidentified IPD will be shared via a secure data transfer mechanism approved by OUHSC. Data sharing requests will be reviewed and approved by the PI and OUHSC.

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT05233228/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT05233228/SAP_001.pdf